CLINICAL TRIAL: NCT02470884
Title: Fully Absorbable Scaffold Feasibility Study
Brief Title: FAST Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2327
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FAST (Experimental): Subjects treated with the Boston Scientific Fully Absorbable Scaffold
  Interventions: Device: Boston Scientific Fully Absorbable Scaffold

INTERVENTIONS:
Device: Boston Scientific Fully Absorbable Scaffold — Attempt to implant the Boston Scientific Fully Absorbable Scaffold.

SUMMARY:
A prospective multi-center, single arm feasibility study to assess the safety and performance of the Boston Scientific Fully Absorbable Scaffold.

DETAILED DESCRIPTION:
The Boston Scientific Fully Absorbable Scaffold is a device/drug combination product providing a mechanical structure for vascular lumen support (the scaffold component) and a pharmacological agent (everolimus) targeted toward reducing the injury response that leads to restenosis after scaffold implantation.

The Boston Scientific Fully Absorbable Scaffold is intended to improve the luminal diameter in subjects with ischemic heart disease due to de novo native coronary artery target lesions ≤ 12 mm in length with reference vessel diameter ≥ 2.75 mm and ≤ 3.25 mm.

Subjects who are candidates for PCI for the treatment of a de novo native coronary artery lesion will be screened according to the protocol inclusion and exclusion criteria. Subjects will be considered enrolled once they have signed the informed consent form and an attempt has been made to implant the fully absorbable study scaffold.

During the index procedure 1 target lesion in a de novo native coronary artery may be treated. Up to 1 non-target lesion in a separate epicardial vessel may be treated with a commercially approved DES

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI) and is an acceptable candidate for coronary artery bypass grafting (CABG)
* Subject has either:

Symptomatic coronary artery disease with one of the following: stenosis > 70%, abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure or Documented silent ischemia based on one of the following: abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure

* Subject is willing to comply with all protocol-required follow-up evaluation
* Target lesion must be <12 mm in length with reference vessel diameter >2.75 mm and <3.25 mm
* Target lesion must have visually estimated stenosis >50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1
* The target lesion must be successfully predilated Note: Successful predilatation refers to dilatation with a balloon catheter of appropriate length and diameter with ≤30% residual stenosis and no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C.

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute MI
* Subjects with unstable angina or recent MI (clinically diagnosed within the past 2 weeks) must have cardiac troponin (cTn) documented prior to the procedure and are excluded if cTn is > 5x ULN
* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
* Non-target vessel or side branch has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to the index procedure
* Target vessel has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 1 year prior to the index procedure
* Planned PCI or CABG after the index procedure
* Subject has a known allergy to contrast that cannot be adequately premedicated or to the study scaffold system or protocol-required concomitant medications (e.g., everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin)
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Subject has a known condition(s) of the following (as assessed prior to the index procedure):

  * Other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Subject previously treated at any time with intravascular brachytherapy
* Subject is receiving chronic (> 72 hours) anticoagulation therapy (i.e., heparin, coumadin) for indications other than acute coronary syndrome
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Subject has a white blood cell (WBC) count <3,000 cells/mm3
* Subject has documented or suspected liver disease that is clinically significant, including laboratory evidence of active hepatitis
* Subject is on dialysis or has baseline serum creatinine level >2.0mg/dL (177µmol/L)
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Subject has signs or symptoms of active heart failure (i.e., is NYHA class IV) at the time of the index procedure
* Subject is participating in another investigational drug or device clinical study that has not reached its primary endpoint
* Subject intends to participate in another investigational drug or device clinical study within 12 months after the index procedure
* Subject is a woman of child-bearing potential with known intention to procreate within 12 months after the index procedure. (Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* Subject is a woman who is pregnant or nursing (A pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
* Planned treatment of more than 1 target lesion and 1 non-target lesion (see below "Multiple Interventions During Index Procedure")
* Planned treatment of the target lesion with more than 1 scaffold
* Target lesion is located in the left main
* Target lesion is located within 3mm of the origin of the left anterior descending (LAD) coronary artery, left circumflex (LCX) coronary artery or right coronary artery (RCA)
* Target lesion is located within a saphenous vein graft or arterial graft or will be accessed via a saphenous vein graft or an arterial graft
* Target lesion involves a side branch >2.0mm in diameter
* Target lesion involves a clinically significant side branch <2.0 mm in diameter that has a clinically significant stenosis at the ostium.
* Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified
* Excessive tortuosity or extreme angulation proximal to or within the target lesion
* Target lesion is restenotic from a previous stent implantation
* Thrombus, or possible thrombus, present in the target vessel
* Non-target lesion to be treated during the index procedure meets any of the following criteria:

  * Located within the target vessel
  * Located within a bypass graft (venous or arterial)
  * Left main location
  * Chronic total occlusion
  * Involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
  * Restenotic from previous intervention
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Clinical Procedural Success | In-hospital (through discharge or 7 days from the index procedure, whichever is sooner)
  Percent diameter stenosis ≤30% and no in-hospital MACE (Death, MI or TLR)

SECONDARY OUTCOMES:
In-scaffold late loss | 6 months
  angiographic endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Sujth Seneviratne, MBBS, Principal Investigator — MonashHeart, Southern Health
Locations (7):
- Australia (4):
  - The Prince Charles Hospital, Chermside, Queensland
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Peninsula Health, Frankston, Victoria
  - Monash Medical Centre, Melbourne, Victoria
- P. Stradins University Hospital, Riga, Latvia
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - North Shore Hospital, Takapuna, Auckland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Outcomes in Patients Treated With the Fully Absorbable, Everolimus-Eluting RENUVIATM Scaffold: Primary Endpoint Results from the FAST First Human Use Study — https://repository.monashhealth.org/monashhealthjspui/handle/1/38998